CLINICAL TRIAL: NCT01826708
Title: Development of a Technique to Identify New Genes by Studying and Cloning the Breakpoints of de Novo Apparently Balanced Chromosomal Translocations in Patients Presenting With Syndromic Psychomotor Retardation
Brief Title: Breakpoint Analysis of de Novo Apparently Balanced Chromosomal Translocations
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UF 8688
Record Dates: First submitted 2012-03-29; First posted 2013-04-08 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2013-04

CONDITIONS: Balanced Chromosomal Translocation
Keywords: Chromosomal translocations; psychomotor delay
MeSH Terms: conditions — Translocation, Genetic; Learning Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Psychomotor retardation syndromic (No Intervention): Psychomotor retardation syndromic by Identification of breakpoints
  Interventions: Biological: Identification of breakpoints

INTERVENTIONS:
Biological: Identification of breakpoints — Identification of breakpoints in Molecular Biology : demonstration of a chimeric sequence corresponding to a junction region between the two chromosomes

SUMMARY:
For every child with developmental delay, the investigators do a constitutional karyotype. This karyotype can reveal an apparently balanced chromosomal rearrangement (no visible loss or gain of genetic material), such as a translocation between two or more chromosomes of accidental occurrence (not transmitted by parents). However, an apparently balanced translocation does not explain the phenotype of the child. Among the hypotheses that could explain the child's symptoms, there is the possibility of another chromosomal abnormality at the translocation breakpoints, another defect elsewhere on the chromosomes or gene disruption at or near the breakpoints. Because the resolution of a constitutional karyotype is limited, these microanomalies can go undiagnosed. The goal of this study is to look for a microanomaly on a chromosome using a technology of higher resolution than that of the conventional karyotype. The proposed study uses DNA microarray technology on DNA extracted from blood lymphocytes to perform high-resolution analysis of all chromosomes to search for an unbalanced microrearrangement (such as loss or gain of chromosomal material). If no microrearrangement is found, the investigators will pursue by looking for a gene disruption defect at or near the breakpoints involved in the translocation. This will be done by first isolating the chromosomes involved in the translocation by flow cytometry and then hybridizing each of the isolated chromosomes on a new microarray. The purpose of this study is to find a possible cause to explain the phenotype (microrearrangement or gene disruption).

DETAILED DESCRIPTION:
Psychomotor delay is observed in approximately 3% of the general population and has various causes: environmental, genetic (gene or chromosome) or unknown. Chromosomal abnormalities have been identified in 15% of syndromic psychomotor delay (ie. associated with another symptom). Balanced chromosomal translocations are observed in one out of every 1000 individuals and only 6% of patients with de novo apparently balanced translocations have an abnormal phenotype (Warburton, 1991). Review of the literature, concerning the microarray analysis of de novo apparently balanced translocations in patients with psychomotor delay, reveals:* in 40% of cases: an abnormality not identified on the karyotype, either at the translocation breakpoints or at a different location on the genome,* in 60% of cases: no abnormalities are found with a resolution of up to 25kb (Schluth-Bolard et al., 2009). The technique generally used to clone a breakpoint and identify a disrupted gene is a "walk" on the chromosome. This technique uses fluorescent probes, such as BACs or PACs, located on the derivative chromosomes on both sides of the breakpoints. This technique is labor-intensive, time-consuming and expensive because one must probe along the derivative chromosomes, closer and closer to the breakpoint, in order to find the probe overlapping the breakpoint. The investigators propose an original, innovative and quick technique to map chromosome translocation breakpoints in patients with psychomotor delay and no abnormalities on microarray analysis. The main aim is to develop a technique to identify new genes by cloning and mapping chromosome translocation breakpoints. These genes would then be candidate to explain the phenotype of the patient.The study covers a 24 month period and includes 10 patients. The feasibility of the technique, as well as its application to routine laboratory diagnosis, will be evaluated. The study was approved by our local Bioethics Committee and respects french law of bioethics.Methodology:Patients well be selected during staff meetings including clinicians and biologists. An initial microarray analysis well be performed to identify a gain or loss of genetic material. Samples for which no gain or loss is identified well then undergo flow cytometry to isolate the derivative chromosomes. Each derivative chromosome well then be hybridised to a new microarray, thus revealing the breakpoint. The breakpoints will be confirmed by FISH technique and molecular biology techniques well be applied to clone and sequence the breakpoints. Databases well be used to check for genes located in or around the breakpoints. Required information: Administrative data (3 first letters of the last name and 2 first letters of the first name, date of birth, identification of parents, informed consent). Clinical and biological data (phenotype, karyotype, other genetic studies). Expected results: Development of rapid and less expensive technique to clone translocation breakpoints, Identification of genes potentially involved in mental delay and anomalies of embryo development, Evaluation of the distribution of various causes of syndromic mental delay (unbalanced translocation on microarray, additional rearrangement on microarray, gene disruption, or unidentified cause).

ELIGIBILITY:
Inclusion Criteria:

* patient with syndromic psychomotor delay
* patient with a apparently balanced de novo chromosomal translocation
* patient with health insurance
* informed consent signed by patient or by parents or by the legal representative for children

Exclusion Criteria:

* patient with an inherited translocation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the proportion of cases for which a cause explaining the phenotype is found for patients with a apparently balance de novo translocation | 6 months and 2 years
  Evaluation of the proportion of cases for which a cause explaining the phenotype is found for patients with a apparently balance de novo translocation

CONTACTS AND LOCATIONS:
Overall Officials: Jacques MD Puechberty, PHD, Principal Investigator — Laboratory of Chromosomal Genetics - Universitary Hospital
Locations (1):
- Laboratory of Chromosomal Genetics - Universitary Hospital, Montpellier, France

REFERENCES:
- [Background] Gribble SM, Prigmore E, Burford DC, Porter KM, Ng BL, Douglas EJ, Fiegler H, Carr P, Kalaitzopoulos D, Clegg S, Sandstrom R, Temple IK, Youings SA, Thomas NS, Dennis NR, Jacobs PA, Crolla JA, Carter NP. The complex nature of constitutional de novo apparently balanced translocations in patients presenting with abnormal phenotypes. J Med Genet. 2005 Jan;42(1):8-16. doi: 10.1136/jmg.2004.024141. PMID 15635069